CLINICAL TRIAL: NCT04311632
Title: A 12-Month, Randomized, Controlled, Open-Label, Dose Escalation Study Evaluating Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of an Anti-CD2 Monoclonal Antibody, TCD601(Siplizumab) Compared to Anti-thymocyte Globulin (rATG), as Induction Therapy in de Novo Renal Transplant Recipients
Brief Title: A Dose Escalation Study in de Novo Renal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TCD601B102
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Tacrolimus; Adrenal Cortex Hormones; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): TCD601 administered with the standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: TCD601; Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF)
- Arm 2 (Experimental): TCD601 administered with the standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: TCD601; Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF)
- Arm 3 (Active Comparator): ATG administered with the standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF); Drug: ATG

INTERVENTIONS:
Biological: TCD601 — Investigational Product
  Arms: Arm 1; Arm 2
Drug: Tacrolimus (TAC) — Standard of Care Concomitant Immunosuppression
Drug: Corticosteroids (CS) — Standard of Care Concomitant Immunosuppression
Drug: Mycophenolate Mofetil (MMF) — Standard of Care Concomitant Immunosuppression
Drug: ATG — Standard of Care induction therapy in solid organ transplantation
  Arms: Arm 3

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of escalating doses of TCD601 when compared to rATG in de novo renal transplant patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand the study requirements and provide written informed consent before and study assessment is performed.
* Male or female patients ≥ 18 to 70 years of age.
* Recipients of a de novo renal allograft from a heart-beating deceased, living unrelated, or non-HLA identical living related donor.
* Recipients of a kidney with a cold ischemia time (CIT) less than 30 hours.

Key Exclusion Criteria:

* Multiple-organ transplant recipients
* Subjects who have received a kidney allograft previously
* Recipient of a kidney from an HLA identical living related donor
* Recipient of a kidney from a donor after cardiac death
* Subjects at high immunological risk for rejection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hryciw, MA, Study Director — ITB-Med LLC
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Barnabas Medical Center, Livingston, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: TCD601 (0.2mg/kg) administered with the standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  TCD601: Investigational Product
  Tacrolimus (TAC): Standard of Care Concomitant Immunosuppression
  Corticosteroids (CS): Standard of Care Concomitant Immunosuppression
  Mycophenolate Mofetil (MMF): Standard of Care Concomitant Immunosuppression
- Arm 2: TCD601 (0.6mg/kg) administered with the standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  TCD601: Investigational Product
  Tacrolimus (TAC): Standard of Care Concomitant Immunosuppression
  Corticosteroids (CS): Standard of Care Concomitant Immunosuppression
  Mycophenolate Mofetil (MMF): Standard of Care Concomitant Immunosuppression
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 2 | 4 | 7
Completed | 2 | 4 | 6
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 2 | 4 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (5.7) | 42 (10.8) | 51.3 (4.7) | 45 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 1 | 4 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 4 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 2 | 3 | 5 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 7 | 13
Height [Mean (Standard Deviation); unit: centimeters] | 171.0 (16.9) | 188.0 (4.4) | 177.7 (8.9) | 179.1 (10.4)
Weight [Mean (Standard Deviation); unit: kilograms] | 66.8 (32.4) | 115.5 (16.5) | 96.8 (19.7) | 97.9 (24.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (6.6) | 30.5 (2.9) | 30.6 (4.6) | 29.0 (5.3)
Viral Serology [Count of Participants; unit: Participants]
  Cytomegalovirus: Positive | 1 | 2 | 3 | 6
  Cytomegalovirus: Negative | 1 | 2 | 4 | 7
  Epstein-Barr Virus: Positive | 2 | 4 | 7 | 13
  Epstein-Barr Virus: Negative | 0 | 0 | 0 | 0
  Hepatitis C Virus Antibody: Positive | 0 | 0 | 0 | 0
  Hepatitis C Virus Antibody: Negative | 2 | 4 | 7 | 13
  Hepatitis B Surface Antigen: Positive | 0 | 0 | 0 | 0
  Hepatitis B Surface Antigen: Negative | 2 | 4 | 7 | 13
  Human Immunodeficiency Virus: Positive | 0 | 0 | 0 | 0
  Human Immunodeficiency Virus: Negative | 2 | 4 | 7 | 13
End Stage Disease Leading to Transplantation [Count of Participants; unit: Participants]
  Glomerular Disease | 1 | 0 | 1 | 2
  Polycystic Disease | 0 | 3 | 0 | 3
  Hypertension/ Nephrosclerosis | 0 | 0 | 2 | 2
  Diabetes Mellitus | 0 | 1 | 3 | 4
  IgA Nephropathy | 0 | 0 | 1 | 1
  Other: Congenital Obstructive Uropathy | 1 | 0 | 0 | 1
Current Dialysis [Count of Participants; unit: Participants]
  Hemodialysis | 0 | 2 | 3 | 5
  Peritoneal Dialysis | 0 | 1 | 2 | 3
  None | 2 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE v5.0.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 2 | 4 | 7
Participants
  At least 1 TEAE: Yes | 2 | 4 | 7
  At least 1 TEAE: No | 0 | 0 | 0
  At least 1 TEAE Related to Study Medication: Yes | 2 | 3 | 4
  At least 1 TEAE Related to Study Medication: No | 0 | 1 | 3
  At least 1 SAE: Yes | 2 | 1 | 5
  At least 1 SAE: No | 0 | 3 | 2
  At least 1 TEAE leading to Study Discontinuation: Yes | 0 | 0 | 0
  At least 1 TEAE leading to Study Discontinuation: No | 2 | 4 | 7
  At least 1 TEAE leading to Dose Adjustment: Yes | 0 | 0 | 0
  At least 1 TEAE leading to Dose Adjustment: No | 2 | 4 | 7
  At least 1 TEAE leading to Dose Interruption: Yes | 0 | 0 | 1
  At least 1 TEAE leading to Dose Interruption: No | 2 | 4 | 6
  At least 1 TEAE leading to Study Medication Discontinuation: Yes | 0 | 0 | 0
  At least 1 TEAE leading to Study Medication Discontinuation: No | 2 | 4 | 7
  At least 1 Infection: Yes | 2 | 3 | 6
  At least 1 Infection: No | 0 | 1 | 1
  At least 1 Serious Infection: Yes | 1 | 0 | 1
  At least 1 Serious Infection: No | 1 | 4 | 6
  At least 1 SAE related to Study Medication: Yes | 1 | 0 | 0
  At least 1 SAE related to Study Medication: No | 1 | 4 | 7

2. Primary Outcome: Measure Peak Plasma Concentration (Cmax) Over Time.
Description: The maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 2 | 4
ug/mL | 5.0 (0.2) | 17.5 (1.1)

3. Primary Outcome: Measure the Area Under the Plasma Concentration Versus Time Curve (AUC).
Description: The AUC from time zero to the last measurable concentration sampling time.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ug/mL*day
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 2 | 4
ug/mL*day | 23.0 (0.5) | 162.0 (53.4)

4. Secondary Outcome: The Incidence of Rejection at 12 Months Post-transplant.
Description: The incidence of treated biopsy-proven acute rejection (tBPAR) and antibody medication rejection (AMR) at 12 months post-transplant.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 2 | 4 | 7
Participants
  tBPAR: Yes | 1 | 0 | 1
  tBPAR: No | 1 | 4 | 6
  AMR: Yes | 0 | 0 | 0
  AMR: No | 2 | 4 | 7

5. Secondary Outcome: To Assess the Change in Renal Function Over Time.
Description: Estimated glomerular filtration rate (eGFR) was calculated using the MDRD4 equation. Mean+-SD eGFR values are presented at 3, 6, and 12. and compared against baseline (1 Month post-transplant).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL/minute/1.73m^2
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 2 | 4 | 7
mL/minute/1.73m^2
  Baseline | 40.4 (5.0) | 50.2 (21.1) | 45.9 (5.8)
  Month 3 | 40.5 (0.3) | 48.2 (9.4) | 48.2 (10.0)
  Month 6 | 39.0 (5.6) | 51.4 (8.9) | 47.2 (17.0)
  Month 12 | 44.0 (7.0) | 53.7 (14.1) | 46.0 (14.3)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/4 | 5/7
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=2) | Arm 2 (N=4) | Arm 3 (N=7)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Perinephric collection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteral necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=2) | Arm 2 (N=4) | Arm 3 (N=7)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (2) | 2 (2) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Polyomavirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Delayed graft function (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
New onset diabetes after transplantation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery dissection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes; and in those instances, the publication shall be resubmitted to the sponsor and will have an additional 30 days for review.

DOCUMENTS (2):
  • Study Protocol (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04311632/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT04311632/SAP_001.pdf